CLINICAL TRIAL: NCT04160221
Title: Second Trimester Medical Abortion- New Strategies
Brief Title: Second Trimester Medical Abortion
Acronym: RAPM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, Dr. Aya Mohr-Sasson, Principal Investigator, Sheba Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6416-19
Record Dates: First submitted 2019-11-06; First posted 2019-11-12 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Medical Abortion, Complete or Unspecified, Without Complication
Keywords: Medical Abortion; Mifepristone; Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 12 hours interval (Active Comparator): Mifepristone followed by Misoprostol treatment
  Interventions: Other: 12 hours interval
- 24 hours interval (Active Comparator): Mifepristone followed by Misoprostol treatment
  Interventions: Other: 24 hours interval

INTERVENTIONS:
Other: 12 hours interval — Time interval between treatments
  Arms: 12 hours interval
Other: 24 hours interval — Time interval between treatments
  Arms: 24 hours interval

SUMMARY:
The use of Mifepristone, an antiprogesterone, and Misoprostol together, has been shown to make the medial abortion process more efficient and reduce the induction-to-abortion interval by almost 50%. Despite the recommended 24-48 Mifepristone-Misoprostol interval, recent retrospective study of a flexible interval, have revealed shorter total abortion time with shorter intervals. In this study we aim to compare 24 to 12 hours Mifepristone to Misoprostol intervals

DETAILED DESCRIPTION:
Women are looking for termination of pregnancies in the second trimester, after 12 weeks of gestation for social and medical reasons, as well as due to intrauterine fetal demise. Both surgical and medical methods can be used, depending on the patients' preference, providers skills, availability of drugs and instruments and more. Methods of medical abortion can be performed with the use of prostaglandin analogues, mifepristone, oxytocin, foley catheter and osmotic dilators. Misoprostol, a prostaglandin analogue (PGE1), is currently recommended over other agents due to its efficacy, low cost and ease of use. Misoprostol can be used alone or in combination with other agents. The use of Mifepristone, an antiprogesterone, and Misoprostol together, has been shown to make the medial abortion process more efficient and reduce the induction-to-abortion interval by almost 50%. Current guidelines recommend the use of Mifepristone 200 mg orally, followed by Misoprostol 400 mcg every 3-4, hours 24-48 later until expulsion of the fetus. Despite the recommended 24-48 Mifepristone-Misoprostol interval, recent retrospective study of a flexible interval, ≤12, 12-24 and >24 hours, have revealed shorter total abortion time (time from Mifepristone to fetal expulsion) with the shorter intervals. Thus, strict adherence to current guidelines may unnecessarily prolong the abortion procedure.

Objective Prompted by the need to explore more beneficial methods and regimes for second trimester medical abortion, we aim to compare 24 to 12 hours Mifepristone to Misoprostol intervals

Material and Methods Women eligible for second trimester medical abortion will be approached to enroll in the study at the clinic or emergency room when they arrive to schedule medical abortion. A research staff member will obtain informed consent. The patient will undergo a blood test including blood type, complete blood count and chemistry. Basic demographic information will be collected. A complete history and physical assessment will be performed. If an ultrasound report is not available to confirm gestational age dating, ultrasound will be performed to determine gestational age. A baseline cervical exam will be done at this visit to assess cervical consistency. Patients will be randomized into one of two groups according to a computer-generated random allocation sequence. Sequentially numbered sealed opaque envelopes will be used to provide allocation.

* Patients allocated to group 1 will receive 200 mg Mifepristone orally, followed by Misoprostol 400 mcg vaginally 12 hours later and subsequently 400 mcg orally every three hours until fetal expulsion to a maximum of 5 doses.
* Patients allocated to group 2 will receive 200 mg Mifepristone orally, followed by Misoprostol 400 mcg vaginally 24 hours later and subsequently 400 mcg orally every three hours until fetal expulsion to a maximum of 5 doses.

Patients will be discharged home after receiving Mifepristone, and hospitalized upon arrival for the Misoprostol administration.

If the abortion is not complete after five doses, the woman may be allowed to rest for 12 hours before starting the cycle again.

All participants will be contacted by phone as well as a chart review conducted to assess for delayed complications. During this follow up time, they will be asked to notify the research team if they should develop fatigue, malaise, abdominal pain, or jaundice. If these symptoms occur, a workup for liver injury would be performed. Patients will be asked to obtain repeat liver function tests within two weeks post-procedure to compare to their baseline hepatic panel.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years and older about to undergo medical second trimester abortion
* 12+0 to 28+0 weeks of gestation
* Singleton intrauterine pregnancy
* Able to sign informed consent

Exclusion Criteria:

* Inability to give informed consent
* Allergy to any of the drugs used in the study
* Genital bleeding of unknown etiology; cancer of the breast, cervix, uterus, or ovaries; hepatic disease (current or history of)
* Multiple gestation
* Rupture of membranes
* Taken a CYP3A4 inhibitor within 5 elimination half-lives of the drug from the procedure
* Pre-dosing abnormal liver function tests
* Patients at increased risk of hepatitis based on a history of any of the following:

  * Any history of underlying liver disorder, including hepatitis
  * A family history of hepatitis or currently living with a person 441 who has been given a diagnosis of hepatitis
  * A history of or currently working as a sex worker
  * A history of or currently using IV drugs
  * A self-reported history of alcoholic dependency or abuse

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 80 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Induction-abortion time | Through completion of abortion, an estimated period of up to 3 days
  Total induction to complete abortion ( estimated by hours)

SECONDARY OUTCOMES:
Fever | From the beginning until completion of abortion,estimated up to two weeks
  Fever measure above 38 degrees
Excessive blood loss | From the beginning until completion of abortion, estimated up to two weeks
  Excessive blood loss estimated by the medical team ( remnants of blood on pad, active bleeding estimated to be equal to menstruation, heavier bleeding including blood clots, blood loss leading to hemodynamically instability including tachycardia and/or reduced blood pressure)
Any emergency department visit | From the beginning until completion of abortion, estimated up to two weeks
  Emergency department visit during the abortion or reported on follow up

CONTACTS AND LOCATIONS:
Overall Officials: Aya A Mohr-Sasson, M.D, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lohr PA, Hayes JL, Gemzell-Danielsson K. Surgical versus medical methods for second trimester induced abortion. Cochrane Database Syst Rev. 2008 Jan 23;(1):CD006714. doi: 10.1002/14651858.CD006714.pub2. PMID 18254113
- [Result] ACOG Practice Bulletin No. 135: Second-trimester abortion. Obstet Gynecol. 2013 Jun;121(6):1394-1406. doi: 10.1097/01.AOG.0000431056.79334.cc. No abstract available. PMID 23812485
- [Result] Borgatta L, Kapp N; Society of Family Planning. Clinical guidelines. Labor induction abortion in the second trimester. Contraception. 2011 Jul;84(1):4-18. doi: 10.1016/j.contraception.2011.02.005. Epub 2011 Mar 30. PMID 21664506
- [Result] Costescu D, Guilbert E. No. 360-Induced Abortion: Surgical Abortion and Second Trimester Medical Methods. J Obstet Gynaecol Can. 2018 Jun;40(6):750-783. doi: 10.1016/j.jogc.2017.12.010. PMID 29861084
- [Result] Li HWR, Gemzell-Danielsson K. Mechanisms of action of emergency contraception pills. Eur J Contracept Reprod Health Care. 2019 Feb;24(1):11-12. doi: 10.1080/13625187.2018.1555663. Epub 2019 Jan 21. No abstract available. PMID 30664367
- [Result] Donnez J, Tomaszewski J, Vazquez F, Bouchard P, Lemieszczuk B, Baro F, Nouri K, Selvaggi L, Sodowski K, Bestel E, Terrill P, Osterloh I, Loumaye E; PEARL II Study Group. Ulipristal acetate versus leuprolide acetate for uterine fibroids. N Engl J Med. 2012 Feb 2;366(5):421-32. doi: 10.1056/NEJMoa1103180. PMID 22296076
- [Result] Blithe DL, Nieman LK, Blye RP, Stratton P, Passaro M. Development of the selective progesterone receptor modulator CDB-2914 for clinical indications. Steroids. 2003 Nov;68(10-13):1013-7. doi: 10.1016/s0039-128x(03)00118-1. PMID 14667994
- [Derived] Meyer R, Toussia-Cohen S, Shats M, Segal O, Mohr-Sasson A, Peretz-Bookstein S, Amitai-Komem D, Sindel O, Levin G, Mashiach R, Blumenthal PD. 24-Hour Compared With 12-Hour Mifepristone-Misoprostol Interval for Second-Trimester Abortion: A Randomized Controlled Trial. Obstet Gynecol. 2024 Jul 1;144(1):60-67. doi: 10.1097/AOG.0000000000005535. Epub 2024 May 23. PMID 38781593